CLINICAL TRIAL: NCT01074567
Title: Efficacy of DMSO Cocktail Treatment in Interstitial Cystitis Patients During and After Treatment
Brief Title: DMSO Efficacy in IC/PBS Patients During and After Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Miki Haifler, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 174/09
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2010-03

CONDITIONS: Cystitis, Interstitial
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMSO cocktail (Experimental): intra-vesical: DMSO 50% in 50 cc water for injection 10 cc heparin 5000 IU hydrocortisone 100 mg bupivacaine 0.125%
  Interventions: Drug: DMSO cocktail

INTERVENTIONS:
Drug: DMSO cocktail — intra-vesical: DMSO 50% in 50 cc water for injection 10 cc heparin 5000 IU hydrocortisone 100 mg bupivacaine 0.125%
  Other Names: Dimethyl sulfoxide

SUMMARY:
The purpose of this study is to examine the efficacy of dimethylsulphoxide (DMSO) cocktail in patients with interstitial cystitis during the treatment period (12 weeks) and after it (at 6 weeks, 3, 6 and 12 month).

DETAILED DESCRIPTION:
The modern treatment of IC is a multi-modal treatment which includes behavioural treatment, physiotherapy of the pelvic floor musculature, oral medication (e.g. Amitryptiline) and intra-vesical instillation (e.g. DMSO, steroids, heparin). These treatments were found to be effective in a number of studies and are approved by the FDA. However, the optimal duration of intra-vesical instilation is not known.

All patients with IC (according to the international continence society criteria) will receive 12 weekly intra-vesical instillation of DMSO. All patients will fill an O'leary-Sant questionaire and a urination diary before treatment, after 3, 6, 9 and 12 treatments and at 6 weeks, 3, 6 and 12 month after the end to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with IC according to International Continence Society:

  * more than 6 month of pelvic pain
  * urinary frequency, urgency, dyspareunia

Exclusion Criteria:

* genitourinary tract infection
* known genitourinary malformation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
O'leary-Sant interstitial cystitis symptom and problem questionaire | before treatment, at 3, 6, 9 and 12 treatments, 6 weeks, 3, 6, 12 month after last treatment

SECONDARY OUTCOMES:
urination diary | before treatment, at 3, 6, 9 and 12 treatments, 6 weeks, 3, 6, 12 month after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf-Harofe MC
Locations (1):
- Assaf Harofe Medical Center, Zeriffin, Israel

REFERENCES:
- See also: international painful bladder foundation — http://www.painful-bladder.org/index.html
- See also: interstitial cystitis association — http://www.ichelp.org